CLINICAL TRIAL: NCT03396081
Title: Efficacy of PRADO Heart Failure in Occitania
Acronym: PRADO-IC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: RECHMPL17_0113; 2017-A01732-51 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2017-12-26; First posted 2018-01-10 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2022-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; Care pathway; Transition program; Efficiency
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRADO-IC (Experimental)
  Interventions: Behavioral: PRADO-IC
- Usual care (Other)
  Interventions: Behavioral: No intervervention Usual Care

INTERVENTIONS:
Behavioral: PRADO-IC — 1. Help of administrative employees to schedule the first medical visits after an hospitalization for heart failure.
  2. Home nurse's visiting program, during 2 to 6 months after the hospitalization for heart failure.
  Arms: PRADO-IC
Behavioral: No intervervention Usual Care — Advices about the care pathway, provided by care givers. Prescription of home nurse's visits if needed.
  Arms: Usual care

SUMMARY:
Patients with heart failure (IC), after hospitalization, have a marked fragility: in France, in the first year, 29% die and 45% are readmitted to IC. Interventions improving the coordination of care providers at the time of discharge from hospitalization were tested; they showed a reduction in readmissions for IC (relative risk (RR) from 0.51 to 0.74) and all-cause mortality (RR 0.75 to 0.87). The Patient Return Program IC (PRADO IC), set up by the Health Insurance, offers assistance in the initiation of outpatient medical monitoring, and a nursing follow-up of 2 to 6 months depending on the patient's severity. The trial of PRADO began in the second half of 2013, and the first evaluation showed that the time to first treatment was significantly shorter, and that the readmissions rate and the 6-month death rate were unchanged.

This study was of epidemiological type, comparative before-elsewhere. The difficulty of controlling for confounders in this type of study limits the scope of these conclusions. The efficacy hypothesis of PRADO IC is therefore always posed in the French context

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Hospitalization for heart failure
* Subject living at home
* Informed consent

Exclusion criteria:

* discharge to a rehabilitation clinic or to medical home for elderly people
* subject without health insurance
* terminal kidney failure
* programmed heart surgery
* waiting for heart transplantation
* psycho-cognitive impairment
* patient not autonomous for mobility at home
* supportive care
* planned move to medical home for elderly people in the coming 6 months
* no fluent french
* not able to provide informed consent
* participating to other study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2022-05-09 (Actual); Study Completion 2022-05-09 (Actual)

PRIMARY OUTCOMES:
Cost-efficacy ratio | 12 months
  Cost to avoid an hospitalization for heart failure

SECONDARY OUTCOMES:
Cost-utility ratio | 12 months
  Cost will be performed from the society perspective. Utility will be derived from the French EQ5D, measured at 0, 6 and 12 months
Number of hospitalization for heart failure | 12 months
  Hospitalizations for heart failure will be defined using claim data.
Number of all causes hospitalization | 12 months
Rate of death from cardiovascular disease | 12 months
Number of general practitionner | 12 months
  Claim data
Number of cardiologist visits | 12 months
  Claim data

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Montpellier, Montpellier, France

REFERENCES:
- [Derived] Roubille F, Labarre JP, Georger F, Galinier M, Herman F, Berdague P, Nogue E, Petroni T, Delbaere Q, Malak A, Robin M, Prunet E, Leclercq F, Pasquie JL, Papinaud L, Mercier G, Ricci JE, Cayla G, Duflos C. PRADOC: A Multicenter Randomized Controlled Trial to Assess the Efficiency of PRADO-IC, a Nationwide Pragmatic Transition Care Management Plan for Hospitalized Patients With Heart Failure in France. J Am Heart Assoc. 2024 Aug 6;13(15):e032931. doi: 10.1161/JAHA.123.032931. Epub 2024 Jul 18. PMID 39023055